CLINICAL TRIAL: NCT04271202
Title: Novel Insight Into Migraine Pathophysiolgy and Galcanezumab Mechanisms of Action
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Rami Burstein, Professor of Anesthesia, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2019P001081
Record Dates: First submitted 2020-02-10; First posted 2020-02-17 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Chronic Migraine
MeSH Terms: interventions — erenumab; galcanezumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Other): Effects of galacenezumab (emgality) treatment (injectable 240 mg initial dose followed by 120 mg treatments 1 and 2 month later) on brain functioning.
  Interventions: Drug: Emgality 120 MG in 1 ML Prefilled Syringe

INTERVENTIONS:
Drug: Emgality 120 MG in 1 ML Prefilled Syringe — Initial dose of 240 mg followed by 2 interventions (1 month apart) of 120 mg - all given as injectables.
  Other Names: Galcanezumab

SUMMARY:
The purpose of this study is to understand better the mechanisms of action of calcitonin gene related peptide (CGRP) targeted monoclonal antibodies in migraine prevention. Specifically, the protocol will allow the investigators to determine whether the main site of action of this novel and recently-approved class of migraine prophylactic drugs act inside or outside the brain and if so, where.

DETAILED DESCRIPTION:
A brief overview of the study: To test the working hypothesis of the study, the investigators propose to study 60 chronic migraine (CM)/high-frequency episodic migraine (HFEM) patients in 4 visits to the Beth Israel Deaconess Medical Center (BIDMC) Comprehensive Headache Center and 2 visits to the imaging center at McLean Hospital. The first 3 visits to BIDMC Comprehensive Headache Center and the first visit to McLean Hospital will take place before treatment, whereas the 4th visit to BIDMC Comprehensive Headache Center and the second visit to McLean Hospital will take place 3 months after initiation of treatment. In these visits, the investigators will collect medical and headache history, perform a physical examination, administer and review subjects' e-diary, and perform functional and structural fMRI brain imaging (see flow chart).

Overall study design: Experimental prospective study involving identification of neurological effects after treatment of CM and HFEM with galcanezumab - an anti-CGRP-monoclonal antibody (mAb).

Design methodologies: Open-label treatment study comparing the effects of galcanezumab on neurological functioning and brain structure in super-responders, responders and non-responders among CM and HFEM patients.

Primary goal: To determine whether galacanezumab - a drug that acts mainly outside the brain - reverses abnormal brain functioning in CM and HFEM patients. For this study, signs of abnormal brain functioning include triggering of migraine by deviation from homeostasis (prodromes, sleep deprivation, skipping meals) and abnormal sensitivity to sensory stimuli (light, noise, smell, auras).

Key details of study implementation: The study includes CM and HFEM patients. The intervention is galacanezumab (Emgality™). Galcanezumab is an anti-CGRP-mAb approved by the FDA for the prophylactic treatment of migraine. Because this is not an efficacy study, the primary endpoint will not include reduction in number of migraine/headache days per month. Rather, the primary endpoints of the study will include the following: incidence of prodromes, incidence of triggers, sensitivity to light, noise and smell during and in between attacks, and incidence of aura (as determined by filling the e-diary), gray mater thickness and connectivity strength between brain areas involved in migraine (as determined by fMRI). Each patient will be scheduled to visit the headache clinic at BIDMC 4 times and the McLean Hospital Pain Imaging Center twice (a total of 6 hospital visits). Visits 1 and 6 (at BIDMC) will take 1 hour. Visits 2 and 4 (at BIDMC) will take 30 min. Visits 3 and 5 (at McLean Hospital) will take 2 hours. In addition, each patient will have to fill a daily diary for 4 months (estimated to take 5 minutes per day), and will receive a 5 minute weekly phone call from a study coordinator.

Participants will undergo the following procedures:

1. Medical and Headache history at BIDMC (questionnaire filled by patients and reviewed by Drs. Ashina and Burstein)
2. Physical examination including measurements of vital signs at BIDMC (performed by Dr. Ashina).
3. E-diary education and administration by study coordinator.

   a. The diary e-diary will be administered in the form of a REDCap survey using an email link that participants can access from their personal computer/electronic device.
4. 2 fMRI sessions at McLean Hospital by Dr. Borsook (see attached protocol from Dr. Borsook at McLean Hospital)
5. Administration of galcanezumab by Dr. Ashina at BIDMC.
6. Self administration of galcanezumab at home

McLean Hospital part of the study: Patients recruited to the study at BIDMC and deemed eligible to participate in the study (per the results of visits 1 and 2), will be referred to McLean Hospital for the fMRI scanning. All fMRI scanning will take place at McLean Hospital under the supervision of our Co-investigator Dr. David Borsook. Subjects will travel to McLean Hospital and be met by the research coordinator at McLean, Jaymin Upadhyay, to escort them to the MRI scanning area. The McLean MRI staff will review the subject's MRI safety checklist and prep the subjects for scanning.Each patient will be scanned twice, once before initiation of treatment with galcanezumab and a second time on day 115 of the study, after being on galcanezumab for about 3 months. Image acquisition will be performed with a Siemens Systems 3 Tesla MRI scanner equipped with a 32-channel head coil. For each patient, a high-resolution, T1-weighted magnetization-prepared rapid gradient-echo sequence will be acquired [slices = 176, field of view = 220 x 220, echo time = 1.74, repetition time = 2520, flip angle = 7°, resolution = 1 x 1 mm, slice thickness = 1 mm, no gap]. Preprocessing for the surface-based morphometric analysis will be performed using FreeSurfer (version 5.3.0) (http://surfer.nmr.mgh.harvard.edu), a semi-automated toolbox for cortical surface reconstruction and visualization Affine registration of the T1-weighted volume to Talairach space is then performed, followed by skull stripping, white matter (WM) segmentation and tessellation of the gray/white matter boundary. Visual inspection and manual correction of topological errors are carried out at each processing step. Following reconstruction of the cortical surface, brains will be inflated, averaged across patients to produce a study-specific brain, and then smoothed using a 10 mm full-width at half maximum Gaussian kernel. Each hemisphere will be parcellated into 34 distinct regions using the Desikan-Killiany atlas. A direct measure of cortical thickness will then be calculated using the shortest distance (mm) between the pial surface and gray-white matter boundary at each point or vertex of the cortical mantle.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 65 years
* Been previously diagnosed with migraine (with or without aura), in accordance with the ICHD-3 (International Classification of Headache Disorders) criteria
* Experiences between 10 to 25 headaches days per month (during the last 3 months), with at least 8 of them being migraine days during which the migraines lasted more than 4 hours if untreated
* Onset of migraine at age 50 years or younger
* Agrees to refrain from initiating or changing the type, dosage, or frequency of any prophylactic medications for indications other than migraine that may interfere with the study objectives (e.g., antidepressants, anticonvulsants, beta-adrenergic blockers, etc.)
* Able to provide written informed consent

Exclusion Criteria:

* Currently on a regimen of 1 or more migraine preventative therapy
* Other significant pain problem (e.g., cancer pain, fibromyalgia, other head or facial pain disorder) that may confound the study assessments
* Known or suspected severe cardiac disease (e.g., symptomatic coronary artery disease, prior myocardial infarction, congestive heart failure)
* Known or suspected cerebrovascular disease (e.g., prior stroke or transient ischemic attack, symptomatic carotid artery disease, prior carotid endarterectomy or other vascular neck surgery)
* Abnormal baseline electrocardiogram (ECG) within the last year (e.g., second or third-degree heart block, prolonged QT interval, atrial fibrillation, atrial flutter, history of ventricular tachycardia or ventricular fibrillation, clinically significant premature ventricular contraction)
* Uncontrolled high blood pressure (systolic >160 mm Hg, diastolic >100 mm Hg) after 3 measurements within 24 hours
* Known history or suspicion of secondary headache
* Known history or suspicion of substance abuse or addiction (within the last 5 years)
* Currently using marijuana (including medical marijuana) or has used marijuana (including medical marijuana) or cannabidiol oil within the last 1 year
* Currently takes simple analgesics or NSAIDs >15 days per month or triptans, ergots, or combined analgesics >10 days per month for headaches or other body pain
* Currently takes prescription opioids for headaches or body pain
* Undergone nerve block (occipital or other) in the head or neck within the last 3 months
* Received botulinum toxin or anti-CGRP-mAb injections within the last 6 months
* Pregnant or thinking of becoming pregnant during the study period, or of childbearing years and unwilling to use an accepted form of birth control
* Participating in any other therapeutic clinical investigation or has participated in a clinical trial in the preceding 30 days
* Belongs to a vulnerable population or has any condition such that his or her ability to provide informed consent, comply with the follow-up requirements, or provide self-assessments is compromised.
* A relative of or an employee of the Investigator or the clinical study site
* Psychiatric or cognitive disorder and/or behavioral problems that, in the opinion of the clinician, may interfere with the study
* History of claustrophobia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-11-22 (Actual)

PRIMARY OUTCOMES:
Change in abnormal brain functioning - sleep deprivation | 1 month before and 3 months after treatment
  Reduction in number of times sleep deprivation (defined as less than 6 hours/night) triggers migraine the next day
Change in abnormal brain functioning - food deprivation | 1 month before and 3 months after treatment
  Reduction in number of times food deprivation (defined as skipping at least 1 meal/day) triggers migraine the same day
Change in abnormal brain functioning - stress | 1 month before and 3 months after treatment
  Reduction in number of times stress (defined by the participant as event that caused temporary stress, such as exam, deadline at work, etc.) triggers migraine the same or next day
Change in abnormal brain functioning - light sensitivity | 1 month before and 3 months after treatment
  Reduction in sensitivity to light (defined as when light intensifies the headache during attacks)
Change in abnormal brain functioning - noise sensitivity | 1 month before and 3 months after treatment
  Reduction in sensitivity to noise (defined as when noise intensifies the headache during attacks)
Change in abnormal brain functioning - smell sensitivity | 1 month before and 3 months after treatment
  Reduction in sensitivity to smell (defined as when smell intensifies and/or triggers the headache)
Change in gray matter volume in the somatosensory cortex | 1 month before and 3 months after treatment
  Measure difference in gray matter volume (as measured in MRI images) in study time frame
Change in BOLD (blood oxygen level-dependent) signal in the visual cortex | 1 month before and 3 months after treatment
  Measure change in BOLD signal (as measured in fMRI images) over study time frame

CONTACTS AND LOCATIONS:
Overall Officials: Rami Burstein, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Pain Clinic at Beth Israel Deaconess Medical Center, Brookline, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ashina S, Melo-Carrillo A, Toluwanimi A, Bolo N, Szabo E, Borsook D, Burstein R. Galcanezumab effects on incidence of headache after occurrence of triggers, premonitory symptoms, and aura in responders, non-responders, super-responders, and super non-responders. J Headache Pain. 2023 Mar 16;24(1):26. doi: 10.1186/s10194-023-01560-x. PMID 36927366